CLINICAL TRIAL: NCT00959920
Title: Study of Obstetric Foley Therapy (SOFT Trial)
Brief Title: Bladder Drainage During Labor: A Randomized Controlled Study of Obstetric Foley Therapy
Acronym: SOFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201539
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Results first posted 2012-05-23 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Labor
Keywords: Indwelling bladder catheter; Intermittent straight catheterization; Labor and Delivery; Time to delivery during labor
MeSH Terms: interventions — Catheters, Indwelling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Indwelling foley catheter (Active Comparator): Insertion of an indwelling foley catheter when bladder emptying is necessary. The indwelling catheter will remain in place until the time of delivery.
  Interventions: Procedure: Indwelling catheter
- Intermittent straight catheterization (Active Comparator): Intermittent straight catheterization will be performed as needed during labor.
  Interventions: Procedure: Intermittent straight catheterization

INTERVENTIONS:
Procedure: Indwelling catheter — Indwelling bladder catheter will remain in place until time of delivery.
  Arms: Indwelling foley catheter
Procedure: Intermittent straight catheterization — intermittent straight catheterization will be performed on an as needed basis until time of delivery.
  Arms: Intermittent straight catheterization

SUMMARY:
The goal of this study is to compare two clinically-relevant bladder drainage techniques. This is a randomized controlled trial with a single primary outcome of time to delivery. The results will inform clinical decisions about method of catheterization during labor.

DETAILED DESCRIPTION:
Urinary catheterization is a common practice during labor following placement of an epidural for pain control, as this form of anesthesia is known to inhibit normal bladder emptying. There is insufficient evidence to guide clinicians in selection of an indwelling catheter versus intermittent straight catheterization during the course of labor.

The goal of this randomized control trial is to compare two clinically-relevant bladder drainage techniques.

ELIGIBILITY:
Inclusion Criteria:

* Women who present to either Loyola University Medical Center or Loyola at Gottlieb Hospital in active labor or for induction of labor with a singleton pregnancy and who are anticipated to undergo vaginal delivery during the current admission

Exclusion Criteria:

* Women who are undergoing a scheduled cesarean delivery
* Women with a contraindication to either of the 2 study interventions
* Multi-fetal gestations
* Current or planned tocolysis
* Women who are on magnesium prophylaxis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarita Massey, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Health System, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rivard C, Awad M, Liebermann M, Dejong M, Massey SM, Sinacore J, Brubaker L. Bladder drainage during labor: a randomized controlled trial. J Obstet Gynaecol Res. 2012 Aug;38(8):1046-51. doi: 10.1111/j.1447-0756.2011.01837.x. Epub 2012 Apr 30. PMID 22540248

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled 7/09-11/09 from the obstetric units of the Loyola University Health System hospitals. Subjects included adult women with a singleton pregnancy who presented to the Labor & Deliver in active labor or for induction, were anticipated to have an normal spontaneous vaginal delivery (NSVD), and had an epidural.
Pre-assignment Details: Every patient was assigned to a group immediately following enrollment.
Period: Overall Study
Arm/Group | Indwelling Foley Catheter | Intermittent Straight Catheterization
Started | 72 | 67
Completed | 72 | 66
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indwelling Foley Catheter | Intermittent Straight Catheterization | Total
Number analyzed (Participants) | 72 | 67 | 139
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 72 | 67 | 139
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (6) | 28.7 (6) | 28.14 (6.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 67 | 139
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 72 | 67 | 139

OUTCOME MEASURES:

1. Primary Outcome: Time to Delivery (by Any Route)
Description: Time to delivery defined as IV placement to delivery of infant.
Time Frame: 1 day
Population: Our a priori sample size required 138 women (69 per group) for 80% power to detect the clinically relevant 30 minute difference in the time to delivery interval with a .05 alpha error.
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Indwelling Foley Catheter | Intermittent Straight Catheterization
Number analyzed (Participants) | 72 | 66
Hours | 10.43 [5.52 to 15.34] | 11.23 [7.15 to 15.31]
Statistical Analysis 1: Comparison: Intermittent Straight Catheterization; The null hypothesis is that patients for whom indwelling foley catheterization was employed will have their time to delivery interval reduced by 30 minutes; Test type: Superiority or Other; p = .42, t-test, 2 sided; Median Difference (Final Values) = .8

2. Secondary Outcome: Difference in Cost Between the Two Interventions
Description: Cost of the intermittent vs. foley catheterization procedures was measured and reported in mean dollars.
Time Frame: End of study.
Population: No formal statistical testing was conducted on these measures as complete financial records were not available for the analysis.
Arm/Group | Indwelling Foley Catheter | Intermittent Straight Catheterization
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Indwelling Foley Catheter | Intermittent Straight Catheterization
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/67
Other Adverse Events (participants affected / at risk) | 0/72 | 0/67

LIMITATIONS AND CAVEATS:
The are not limitations or caveats to disclose.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes